CLINICAL TRIAL: NCT00283699
Title: A Pilot Study of Neurocysticercosis Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: W Allen Hauser, Professor of Neurology and Epidemiology, College of Physicians and Surgeons and Mailman School of Public Health, Columbia University
Organization: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01NS039403 (NIH)
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2008-03

CONDITIONS: Neurocysticercosis
Keywords: neurocysticercosis; albendazole; tape worm
MeSH Terms: conditions — Neurocysticercosis | interventions — Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 1. albendazole, 15 mg/kg/day for those less than 50 kg in weight. For those more than 50 kg, 800 mg was administered. All got standard symptomatic therapy
  2. placebo plus standard symptomatic therapy
  Interventions: Drug: albendazole
- 2 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: albendazole — Active drug or placebo dosed bid p o for 8days
  Arms: 1
Other: placebo — an inactive substance
  Arms: 2

SUMMARY:
The purpose of this study is to determine if treatment with albendazole improves the clinical outcome of neurocysticercosis infection and/or leads to the disappearance of cysts sooner when compared with symptomatic treatment.

DETAILED DESCRIPTION:
Neurocysticercosis-a disease in which a young tapeworm infects the brain-is common in much of the developing world. It affects approximately 1 out of every 10 people in the United States and is said to be the primary cause of adult-onset epilepsy. The infection creates cysts in the brain, causing seizures and headaches among other symptoms. To date no successful preventive treatment for neurocysticercosis exists.

At present, medicines that kill the adult tapeworm in the stomach and intestines are also used to treat neurocysticercosis caused by the young tapeworm. However, in cases of neurocysticercosis, the methods of administration, doses, and duration of treatment with these medicines still have not been determined. Although these medicines may kill the worm in the brain more rapidly than the natural mechanisms of the body, the long-term benefit of using the medicines to eliminate the worms after the first 1 or 2 months is not clear. In addition, the drugs that kill the worm may be associated with in increased seizures and headache during treatment, and may cause inflammation of the meninges-the covering of the brain-leading to symptoms that may require surgery.

The goal of this trial is to determine if treatment with the antiparasitic agent albendazole improves the outcome of neurocysticercosis infection. This trial will also determine if albendazole leads to the disappearance of cysts sooner when compared with symptomatic treatment.

Participants will be randomly assigned to receive either the study medication, albendazol, or a placebo, an inactive substance, for an 8-day inpatient or outpatient therapy period. Additionally, all participants will receive prednisolone, a corticosteroid, as well as other medications. Participants will remain under the care of a doctor for 2 years and will have regularly scheduled visits and testing.

Information learned in this study may lead to improved treatment of neurocysticercosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with new onset of symptoms associated with neurocysticercosis within two months of identification and have active and/or transitional neurocysticercosis cysts on computed tomography (CT) or magnetic resonance imaging (MRI)

Exclusion Criteria:

* Patients with only calcifications
* Patients who are pregnant
* Patients with one of the following conditions: papilledema, active tuberculosis, syphilis, ocular cysticercosis, active gastric ulcers, or a progressive and life-threatening disorder
* Patients who received anthelmintic drugs (AHD) during the year preceding presentation or who received steroids within 30 days of presentation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2001-02; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Cyst freedom | 1 month, 6 months, 1 year

SECONDARY OUTCOMES:
cyst reduction | 1 month, 6 months, 1 year
seizure freedom | actuarial at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: W. Allen Hauser, MD, Principal Investigator — G.H. Sergievsky Center, Columbia University
Locations (5):
- Ecuador (5):
  - Vicente Corral Moscoso Hospital of Cuenca, Centro de Epilepsia, Facultad de Ciencias Médicinas de la Universidad de Cuenca IDIUC (Área 5), Av. 12 de Abril. Cdla., Cuenca
  - Teodoro Maldonado Carbo Hospital, Av. 25 de Julio Vía Puerto Marítimo, Guayaquil
  - Baca Ortiz Children's Hospital, Av. Colon s/n y 6 de Diciembre, Quito
  - Hospital Carlos Andrade Marin, Av. 10 de agosto y Bogotá, Quito
  - Hospital Eugenio Espejo, Servicio de Neurología, Av. Colombia s/n, Quito

REFERENCES:
- [Derived] Carpio A, Kelvin EA, Bagiella E, Leslie D, Leon P, Andrews H, Hauser WA; Ecuadorian Neurocysticercosis Group. Effects of albendazole treatment on neurocysticercosis: a randomised controlled trial. J Neurol Neurosurg Psychiatry. 2008 Sep;79(9):1050-5. doi: 10.1136/jnnp.2008.144899. Epub 2008 May 21. PMID 18495737